CLINICAL TRIAL: NCT02247323
Title: Ovarian Malignancy Incidence in Premenopausal Women Who Were at Moderate Risk for Malignancy by Risk of Malignancy Index With Low CA 125.(Retrospective Study)
Brief Title: Ovarian Malignancy Incidence in Moderate Risk Women With Low CA 125
Acronym: CA125
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Assistant Professor of Obstetrics and Gynecology, Beni-Suef University
Other Study IDs: Beni-Suef 6
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- premenopausal women: premenopausal women with complex ovarian mass moderate for malignancy by risk of malignancy index score and low CA125.
  Interventions: Other: Risk of malignancy index

INTERVENTIONS:
Other: Risk of malignancy index — Calculation of RMI before sugery.
  Other Names: RMI

SUMMARY:
The investigators are assessing the incidence of ovarian cancer in premenopausal women who were at moderate risk of malignancy with low CA125.

DETAILED DESCRIPTION:
About 10% of premenopausal women may have a surgery for ovarian masses. In premenopausal women the incidence of ovarian malignancy is 1:1000 in case of symptomatic ovarian cyst.1 CA125 is unreliable in differentiating benign from malignant ovarian mass in premenopausal women due to many false positive results and reduced specificity.1 pelvic vaginal ultrasonography is the most effective tool in evaluating ovarian masses due to increased sensitivity over abdominal US.1 An estimation of risk of malignancy index is essential in evaluating an ovarian mass.26 /2 Risk of malignancy index combines presurgical features serum including CA125, menopausal status and ultrasound findings. RMI=Ux Mx CA125 in which each feature takes a score and after calculation score less than 25 is mild, from 25-250 moderate and more than 250 has a severe risk of malignancy needing oncologist.44/3

ELIGIBILITY:
Inclusion Criteria:

* Women with complex ovarian cyst
* Abdominal pain
* Menometrorrhagia

Exclusion Criteria:

* Significant weight loss
* Cachexia
* History of ovarian or other malignancy
* Family history of ovarian Cancer

Ages: 45 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal who had complex ovarian mass with low CA125 and at moderate risk for malignancy by RMI.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of ovarian malignancy | one year
  Calculation of number of women who had ovarian cancer after an operation in moderate risk

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen A Shehata, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University, Cairo, Egypt

REFERENCES:
- See also: National Institute for health and clinical excellence. Ovarian cancer:The recognition and initial management of ovarian cancer.NICE clinical guideline 122.London:NICE;2011 — http://www.google.com.eg/search?q=National+Institute+for+health+and+clinical+excellence.+Ovarian+cancer%3AThe+recognition+and+initial+management+of+ovarian+cancer.NICE+clinical+guideline+122.London%3ANICE%3B2011&oq=National+In